CLINICAL TRIAL: NCT03983044
Title: Comparison of Two Methods for Assessing Cough Capacity in Intensive Care Unit After Cardiac Surgery: Parietal Ultrasound vs. Peak Expiratory Cough Flow
Brief Title: Comparison of Two Methods for Assessing Cough Capacity in Intensive Care Unit After Cardiac Surgery
Acronym: DEPT
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01114-51
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-05

CONDITIONS: Intensive Care Unit; Cardiac Surgery
Keywords: cough evaluation; intensive care unit; utrasound evaluation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Weaning from mechanical ventilation represents 50% of the time spent under mechanical ventilation (1). The risk factors identified in the failure to wean from mechanical ventilation are:

* left heart dysfunction with LVEF < 30%.
* an ineffective cough
* presence of resuscitation neuromyopathy
* mechanical ventilation time >7 days
* presence of a delirium
* age >65 years old
* abundant bronchial secretion
* presence of underlying lung pathology An ineffective cough is found in 40% of patients requiring reintubation. However, cough assessment is most often approximate, based on a subjective assessment of cough strength by asking the patient to cough spontaneously on his or her tube).

The objective evaluation of cough is based on the measurement of the peak expiratory flow rate at cough, commonly referred to as peak expiratory flow rate at cough (PEFD), the patient is asked to take a deep breath and then cough as hard as possible.

Subjective cough assessment does not predict the occurrence of ventilatory withdrawal failure. Conversely, all studies that objectively assessed the strength of cough before extubation by measuring the PEFD found a significant association with the outcome of extubation: a low PEFD increases the risk of extubation failure by a factor of 5 to 9.

The investigators hypothesize that the increase in parietal abdominal muscle contraction obtained by using a non-invasive ultrasound method indicates an effective cough. Conversely, an ineffective cough can be detected by this simple ultrasound criterion, which can be performed at the patient's bedside and extrapolated to all intensive care units equipped with an ultrasound scanner. This evaluation will be carried out before extubation: during the spontaneous ventilation test on a tube in a half-seated position (>45°) and within 24 hours after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Major patients admitted for intubated resuscitation, ventilated after sternotomy cardiac surgery and having a mechanical ventilation time of less than 48 hours.

Exclusion Criteria:

* Pregnant patient
* Recent history of stroke(<6 months )
* Minor patient
* Neurological disorder (Alzheimer's disease, delirium, confusion)
* Emphysemal patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to intensive care, intubated after cardiac surgery by sternotomy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
parietal ultrasound | 48 hours
  compare parietal ultrasound with peak expiratory flow rate measurement (PEFD) in patients ventilated less than 48 hours after cardiac surgery with a sternal approach.
peak expiratory flow rate | 48 hours
  compare parietal ultrasound with peak expiratory flow rate measurement (PEFD) in patients ventilated less than 48 hours after cardiac surgery with a sternal approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No